CLINICAL TRIAL: NCT01238029
Title: Combinational Therapy of Capecitabine, Lapatinib and Vinorelbine for the Treatment of Patients With her2/Neu Positive, Relapsed or Metastatic Breast Carcinoma Following Treatment Failure With Trastuzumab
Brief Title: Dose Finding Study for Combination of Capecitabine, Lapatinib and Vinorelbine in Metastatic Breast Cancer
Acronym: CELAVIE
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: new methods of treatment, no more patients appilicable for study
Sponsor: Sponsor GmbH (Other)
Collaborators: iOMEDICO AG (Industry); Arbeitsgemeinschaft fur Internistische Onkologie (Other); Arbeitskreis Klinische Studien (Other); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0907-002
Record Dates: First submitted 2010-11-02; First posted 2010-11-10 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Metastatic Breast Cancer; HER2 Positive; First or Second Line Therapy; Failure or Contraindication of Trastuzumab Therapy
Keywords: Dose finding study; Combination
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib; Capecitabine; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Capecitabine, Lapatinib, Vinorelbine (Experimental)
  Interventions: Drug: Lapatinib and Capecitabine and Vinorelbine

INTERVENTIONS:
Drug: Lapatinib and Capecitabine and Vinorelbine — Dose finding Study Lapatinib: 1000-1250 oral, once daily, days 1-21 Capecitabine: 1000 mg/sqm oral, bid, days 1-14 Vinorelbine 10-22,5 mg/sqm, i.v. Day 1 + 8
  Other Names: Xeloda; Tyverb; Navirel

SUMMARY:
The purpose of the study is to investigate safety and efficiency of the triple combination of capecitabine, lapatinib and vinorelbine in patients with metastatic breast cancer.

DETAILED DESCRIPTION:
The combination of lapatinib with capecitabine ist a standard therapy für Her2 positive metastatic breast cancer. This study combines this therapy with the additional antimitotic mode of function by vinorelbine.

ELIGIBILITY:
Key Inclusion Criteria:

* Written informed consent
* Able to comply with the protocol
* ECOG performance status 0-1
* Adequate contraception
* Confirmed Her2/neu-positive, adenocarcinoma of the breast
* At least one measurable lesion according to RECIST 1.1 criteria
* First or second chemotherapy after diagnosis of metastasis
* Lapatinib treatment indicated (adjuvant trastuzumab treatment <12 months ago or progressive disease with trastuzumab treatment)
* No signs and symptoms of CHF (chronic heart failure), LVEF (left ventricular ejection fraction) at study start at least 55%
* Adequate hepatic and renal function value
* Adequate hematologic function values

Exclusion Criteria:

* Pregnant or lactating women
* Concurrent participation in another clinical trial. Prior participation is allowed if the last study medication was administered more than 4 weeks prior to randomization
* Asymptomatic with regards to tumor illness
* Previous treatment with lapatinib, capecitabine or vinorelbine
* Necessity of planned treatment with other chemotherapeutics oder anti-hormone therapy
* Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to randomization, or anticipation of the need for major surgery during the course of the study
* Evidence of cardiovascular disease, e.g. myocardial infection, unstable angina pectoris or arrhythmia
* History of vascular or cardiovascular disease within the past 6 months
* All illnesses that result in malabsorption of oral medication or inability to take oral medication
* Concurrent treatment with anti-viral drugs based on sorivudine or with aminoglycosides
* Concurrent treatment with any drug interfering with study medication, especially, those that induce CYP3A
* Concurrent treatment with allopurinol
* Other malignancies (except for basal cell carcinoma of the skin and cervical carcinoma in situ); patient can be included in the study if no recurrent disease has been observed for at least 5 years
* Concurrent illnesses or other circumstances that could interfere with trial participation, efficacy or safety of the patient

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-10; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Identification of maximal tolerable Dose (MTD) of combination with Capecitabine and Lapatinib and Vinorelbine | 4 months
  Phase I: Identification of Dosis limiting toxicities and maximal tolerable dose for Combinational therapy (Time Frame: within the first 21 days under medication)

SECONDARY OUTCOMES:
Overall response Rate | 12 months
  Measurement with CT or MRI after three and six cycles and every three months, as long no tumor progression is detected.
Progression free survival | 12 months
  Measurement with CT or MRI after three and six cycles and every three months, as long no tumor progression is detected.
Time to treatment failure (TTF) | 12 months
  Measurement with CT or MRI after three and six cycles and every three months, as long no tumor progression is detected.
Overall survival (OS) | 12 months
  Measurement with CT or MRI after three and six cycles and every three months, as long no tumor progression is detected.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Soeling, MD, Principal Investigator — Goethestr. 47, 34119 , Kassel, Germany
Locations (11):
- Germany (11):
  - Onkologie Ravensburg, Ravensburg, Baden-Wurttemberg
  - Praxisgemeinschaft Dres. Siehl und Söling, Kassel, Hesse
  - Onkologische Schwerpunktpraxis, Goslar, Lower Saxony
  - Onkologische Schwerpunktpraxis Leer Emden, Leer, Lower Saxony
  - Schwerpunktpraxis Hämatologie / Onkologie, Stade, Lower Saxony
  - Onkodok (Dr. Rösel und Dr. Depenbusch), Gütersloh, North Rhine-Westphalia
  - Praxis für Hämatologie und Onkologie, Mülheim, North Rhine-Westphalia
  - Hämatologisch-onkologische Gemeinschaftspraxis, Münster, North Rhine-Westphalia
  - Praxis für Onkologie u. Hämatologie, Neuss, North Rhine-Westphalia
  - Onkologische Gemeinschaftspraxis Dörfel/Göhler, Dresden, Saxony
  - Onkologische Schwerpunktpraxis, Heidelberg